CLINICAL TRIAL: NCT00946712
Title: A Randomized, Phase III Study Comparing Carboplatin/Paclitaxel or Carboplatin/Paclitaxel/Bevacizumab With or Without Concurrent Cetuximab in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: S0819: Carboplatin and Paclitaxel With or Without Bevacizumab and/or Cetuximab in Treating Patients With Stage IV or Recurrent Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated at pre-planned futility analysis
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0819; NCI-2009-01664 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000649817; S0819 (Other: SWOG); S0819 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Large Cell Lung Carcinoma; Recurrent Lung Adenocarcinoma; Recurrent Squamous Cell Lung Carcinoma; Stage IV Large Cell Lung Carcinoma; Stage IV Lung Adenocarcinoma; Stage IV Squamous Cell Lung Carcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Cetuximab; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (chemo +/- bevacizumab) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes with or without bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients receiving bevacizumab may continue to receive bevacizumab (as above) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (chemo, cetuximab, +/- bevacizumab) (Experimental): Patients receive paclitaxel and carboplatin with or without bevacizumab as in Arm I. Patients also receive cetuximab IV over 1-2 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients may continue to receive cetuximab with or without bevacizumab (as above) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Biological: Cetuximab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm II (chemo, cetuximab, +/- bevacizumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This randomized phase III trial studies carboplatin and paclitaxel to compare how well they work with or without bevacizumab and/or cetuximab in treating patients with stage IV or non-small cell lung cancer that has returned after a period of improvement (recurrent). Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab may prevent the growth of new blood vessels that tumor needs to grow. Cetuximab may also stop cancer cells from growing by binding and interfering with a protein on the surface of the tumor cell that is needed for tumor growth. It is not yet known whether giving carboplatin and paclitaxel are more effective with or without bevacizumab and/or cetuximab in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival (OS) in the entire study population. II. To compare progression-free survival (PFS) by institutional review of epidermal growth factor receptor (EGFR) fluorescent in situ hybridization (FISH)-positive patients.

SECONDARY OBJECTIVES:

I. To compare OS and PFS by centralized review in EGFR FISH-positive patients. II. To compare PFS by centralized image review and by institutional review in the entire study population.

III. To compare the response rate (confirmed plus unconfirmed, complete and partial responses) in a subset of patients with measurable disease in EGFR FISH-positive patient and the entire study population.

IV. To assess the toxicities of these treatment regimens. V. To prospectively test EGFR FISH as a predictive marker for the selection of patients for cetuximab plus chemotherapy.

III. To evaluate the role of V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) mutations in terms of cetuximab efficacy.

IV. To compare the results of EGFR FISH with KRAS mutations, EGFR mutations, EGFR immunohistochemistry (IHC), and other purported EGFR-related biomarkers.

TERTIARY OBJECTIVES:

I. To compare PFS in patients with advanced non-small cell lung cancer (NSCLC) with an IHC score > 200 treated with carboplatin, paclitaxel, and bevacizumab (if appropriate) with or without cetuximab.

II. To compare OS in patients with advanced NSCLC with an IHC score > 200 treated with carboplatin, paclitaxel, and bevacizumab (if appropriate) with or without cetuximab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes with or without bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients receiving bevacizumab may continue to receive bevacizumab (as above) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel and carboplatin with or without bevacizumab as in Arm I. Patients also receive cetuximab IV over 1-2 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, patients may continue to receive cetuximab with or without bevacizumab (as above) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven primary non-small cell lung cancer (adenocarcinoma, large cell carcinoma, squamous or unspecified); disease must be stage IV; disease may be either newly diagnosed or recurrent after previous surgery and/or irradiation; patients with additional lesions in an ipsilateral non-primary lobe without M1a or M1b disease will not be considered to have stage IV disease and are not eligible
* Patients must have a computed tomography (CT) or magnetic resonance imaging (MRI) scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to registration; patient must not have brain metastases unless: (1) metastases have been treated and have remained controlled for at least two weeks following treatment, AND (2) patient has no residual neurological dysfunction off corticosteroids for at least 1 day
* Patients may have measurable or non-measurable disease documented by CT or MRI; the CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality; measurable disease must be assessed within 28 days prior to registration; pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease; non-measurable disease must be assessed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients must have tumor tissue available for submission that is sufficient for EGFR FISH testing and must agree to submission of these specimens; patients must also agree to submission of specimens for other translational medicine studies; patient must be offered participation in banking for future research
* Patients must not have received prior chemotherapy for any stage non-small cell lung cancer; patients must not have received prior platinum-based chemotherapy for any purpose; patient must not have received any cetuximab, gefitinib, erlotinib, or other investigational agents that target the EGFR pathway; patients must not have received for any purpose prior bevacizumab or other vascular endothelial growth factor (VEGF)-related agents; patients must not have received for any purpose prior chimerized or murine monoclonal antibody therapy or have documented presence of human anti-mouse antibodies (HAMA)
* Prior radiation is permitted; however, patients must have recovered from all associated toxicities at time of registration; in order to qualify as measurable, measurable disease must be outside the previous radiation field or must have progressed
* Time from surgical or biopsy procedures is dependent on whether it is planned for the patient to receive bevacizumab

  * For patients who are bevacizumab-appropriate AND bevacizumab is planned: at least 28 days must have elapsed since major surgery (i.e. thoracotomy or video-assisted thoracoscopic surgery [VATS] resection of lung cancer, open pleural biopsy or another major surgical procedure such as abdominal surgery) or significant traumatic injury; patients must have recovered from all associated toxicities at the time of registration; there must be no anticipation of need for major surgical procedures during protocol treatment; patients must not have had a core biopsy, mediastinoscopy, pleurodesis, VATS pleural biopsy or VATS pericardial window within 14 days prior to registration; patients must not have had a percutaneous fine needle aspiration (FNA), thoracentesis or central venous access device implanted within 7 days prior to registration; for other surgical procedures not listed here, please contact the study coordinators
  * For patients who are bevacizumab-inappropriate or bevacizumab is not planned: at least 28 days must have elapsed since major surgery (i.e. thoracotomy or VATS resection of lung cancer, open pleural biopsy or another major surgical procedure such as abdominal surgery) or significant traumatic injury; patients must have recovered from all associated toxicities at the time of registration; there must be no anticipation of need for major surgical procedures during protocol treatment; patients must not have had a core biopsy, mediastinoscopy, pleurodesis, VATS pleural biopsy or VATS pericardial window within 7 days prior to registration; patients must not have had a percutaneous fine needle aspiration (FNA), or thoracentesis within 1 day prior to registration; patients may have had a central venous access device placed at any time prior to registration; for other surgical procedures not listed here, please contact the study coordinators
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Hemoglobin >= 9 g/dL
* Serum creatinine =< institutional upper limit of normal (IULN) AND calculated or measured creatinine clearance >= 50 cc/min using the following Cockroft-Gault formula
* For patients who will be receiving bevacizumab, urine protein must be screened by urine analysis for urine protein creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein must be obtained and the level must be < 1,000 mg for patient enrollment; the urine protein used to calculate the UPC ratio must be obtained within 14 days prior to registration; UPC or 24-hour protein is not required for patients who will not receive bevacizumab Note: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* Serum bilirubin =< 2 times IULN (for patients with liver metastases, bilirubin must be =< 5 X IULN)
* Serum glutamic oxaloacetic transaminase (SGOT) OR serum glutamate pyruvate transaminase (SGPT) =< 2 times IULN (for patients with liver metastases, either SGOT or SGPT must be =< 5 X IULN)
* Zubrod performance status 0-1
* Patients must not have >= grade 2 symptomatic neuropathy-sensory (National Cancer Institute [NCI] Common Terminology Criteria version 3.0)
* Patients must not have documented evidence of acute hepatitis or have an active or uncontrolled infection
* Patients must not have the following: history (within past 6 months) of cerebrovascular accident (CVA), myocardial infarction or unstable angina; or at the time of registration, uncontrolled hypertension, New York Heart Association grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or clinically significant peripheral vascular disease
* Patients must have no known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies (examples include trastuzumab [Herceptin] and epoetin alpha)
* Patients must be willing to provide prior smoking history
* No other prior malignancy is allowed except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1333 (Actual)
Dates: Start 2009-07-15; Primary Completion 2017-08-31 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Herbst, Principal Investigator — SWOG Cancer Research Network
Locations (798):
- United States (797):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Gulf Coast MBCCOP, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - The University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Medical Oncology Hematology Medical Associates-Antioch, Antioch, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Enloe Medical Center, Chico, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Northbay Cancer Center, Fairfield, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mather Veteran Affairs Medical Center, Mather, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Diablo Valley Oncology and Hematology Medical Group-Pleasant Hill, Pleasant Hill, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - East Bay Medical Oncology Hematology Associates Inc, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Saint Helena Hospital, St. Helena, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Denver Veterans Administration Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Bayhealth Medical Center at Kent General, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Gainesville Hematology Oncology Associates, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sacred Heart Medical Oncology Group - Davis Highway, Pensacola, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Resurrection Healthcare, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Central Illinois CCOP, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Galesburg Cottage Plaza Office, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Cadence Cancer Center at Delnor, Geneva, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Center-West, Kansas City, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center-Shawnee Mission, Shawnee Mission, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Caritas Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren-Bay Region, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Great Lakes Cancer Institute, Clarkston, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Great Lakes Cancer Institute-Lapeer Campus, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - McLaren-Macomb, Mount Clemens, Michigan
  - McLaren-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Forest General Hospital, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Christian Hospital Northeast - Northwest, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Sunrise, Las Vegas, Nevada
  - Children's Specialty Center of Nevada II, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Reno Oncology Consultants, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Kennedy Health Systems-Cancer Center, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Coney Island Hospital, Brooklyn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Carolinas Medical Center-Union, Monroe, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Regional Medical Center, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Cancer Control Consortium CCOP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology and Hematology Care Inc-Taft, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Oncology Inc, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Surgical Associates Inc, Tulsa, Oklahoma
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Saint Charles Medical Center-Bend, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Riddle Hospital, Media, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Mercy Suburban Hospital and Cancer Center, Norristown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Mercy Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology-Austin North, Austin, Texas
  - Texas Oncology-Cedar Park, Cedar Park, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology- San Marcos, San Marcos, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Auburn Regional Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative of Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Instituto Nacional De Cancerologia de Mexico, Tlalpan, Mexico

REFERENCES:
- [Derived] Hirsch FR, Redman MW, Moon J, Agustoni F, Herbst RS, Semrad TJ, Varella-Garcia M, Rivard CJ, Kelly K, Gandara DR, Mack PC. EGFR High Copy Number Together With High EGFR Protein Expression Predicts Improved Outcome for Cetuximab-based Therapy in Squamous Cell Lung Cancer: Analysis From SWOG S0819, a Phase III Trial of Chemotherapy With or Without Cetuximab in Advanced NSCLC. Clin Lung Cancer. 2022 Jan;23(1):60-71. doi: 10.1016/j.cllc.2021.10.002. Epub 2021 Oct 10. PMID 34753703
- [Derived] Herbst RS, Redman MW, Kim ES, Semrad TJ, Bazhenova L, Masters G, Oettel K, Guaglianone P, Reynolds C, Karnad A, Arnold SM, Varella-Garcia M, Moon J, Mack PC, Blanke CD, Hirsch FR, Kelly K, Gandara DR. Cetuximab plus carboplatin and paclitaxel with or without bevacizumab versus carboplatin and paclitaxel with or without bevacizumab in advanced NSCLC (SWOG S0819): a randomised, phase 3 study. Lancet Oncol. 2018 Jan;19(1):101-114. doi: 10.1016/S1470-2045(17)30694-0. Epub 2017 Nov 20. PMID 29169877
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Started | 671 | 662
Completed | 124 | 0
Not Completed | 547 | 662
Not completed — Adverse Event | 118 | 124
Not completed — Disease progression | 308 | 404
Not completed — Death | 21 | 22
Not completed — No treatment given | 25 | 29
Not completed — Other reasons | 61 | 73
Not completed — On Treatment | 0 | 4
Not completed — Ineligible | 14 | 6

BASELINE CHARACTERISTICS:
Population: Only eligible patients are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab) | Total
Number analyzed (Participants) | 657 | 656 | 1313
Age, Continuous [Median (Full Range); unit: years] | 63 [30 to 86] | 63 [19 to 84] | 63 [19 to 86]
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorized: Age <= 65 | 379 | 381 | 760
  Age, Categorized: Age > 65 | 278 | 275 | 553
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 271 | 569
  Male | 359 | 385 | 744
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 16 | 42
  Not Hispanic or Latino | 606 | 618 | 1224
  Unknown or Not Reported | 25 | 22 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 565 | 568 | 1133
  Race: Black | 61 | 55 | 116
  Race: Asian | 10 | 18 | 28
  Race: Pacific Islander | 3 | 6 | 9
  Race: Native American | 2 | 1 | 3
  Race: Unknown | 16 | 8 | 24
M-stage [Count of Participants; unit: Participants] — M staging per AJCC Cancer Staging Manual, 7th Edition, 2009. M1a: Separate tumor nodule(s) in a contralateral lobe; tumor with pleural nodules or malignant pleural (or pericardial) effusion.
  M1b: Distant metastases
  Participants
    M1a | 148 | 150 | 298
    M1b | 509 | 506 | 1015
Bevacizumab treatment [Count of Participants; unit: Participants]
  Yes | 277 | 283 | 560
  No | 380 | 373 | 753
Smoking History [Count of Participants; unit: Participants]
  Current | 297 | 292 | 589
  Former | 303 | 305 | 608
  Never | 57 | 59 | 116
Histology [Count of Participants; unit: Participants] — 'Other' includes large-cell carcinoma, bronchioloalveolar carcinoma, mixed, other, and not reported.
  Participants
    Squamous cell carcinoma | 161 | 160 | 321
    Adenocarcinoma | 408 | 411 | 819
    Other | 88 | 85 | 173
Performance Status [Count of Participants; unit: Participants] — Patients will be graded according to the Zubrod Performance Status Scale. 0 Fully active, able to carry on all pre-disease performance without restriction.
  1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 229 | 256 | 485
    1 | 427 | 400 | 827
    Missing Data | 1 | 0 | 1
EGFR (Epidermal Growth Factor Receptor) FISH (Fluorescence In Situ Hybridization) status [Count of Participants; unit: Participants]
  Positive | 201 | 199 | 400
  Negative | 293 | 283 | 576
  Unknown | 163 | 174 | 337

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the Entire Study Population
Description: From date of randomization to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Patients will be followed every 3 weeks while on protocol treatment. Once off all protocol treatment, patients will be followed every 6 months until death or up to 3 years
Population: All eligible patients are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 657 | 656
months | 9.2 [8.7 to 10.3] | 10.9 [9.5 to 12.0]
Statistical Analysis 1: Comparison: Arm I (Chemo +/- Bevacizumab) vs Arm II (Chemo, Cetuximab, +/- Bevacizumab); Test type: Other; p = 0.22, Log Rank; A stratified log rank test was used; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.83 to 1.04]

2. Primary Outcome: Progression-free Survival (PFS) of EGFR FISH-positive Patients by Institutional Review
Description: From date of randomization to date of first documentation of progression or symptomatic deterioration, or death due to any cause, whichever comes first by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as assessed by the treating investigator.Patients last known to be alive and progression-free are censored at date of last contact. Progression is defined using RECIST 1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Disease assessment will be repeated every 6 weeks for the first 9 months and every 3 months thereafter, until disease progression.
Population: Eligible patients with EGFR FISH positive are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 201 | 199
months | 4.8 [3.9 to 5.5] | 5.4 [4.5 to 5.7]
Statistical Analysis 1: Comparison: Arm I (Chemo +/- Bevacizumab) vs Arm II (Chemo, Cetuximab, +/- Bevacizumab); Test type: Other; p = 0.40, Log Rank; A stratified log rank test was used; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.75 to 1.12]

3. Secondary Outcome: Overall Survival (OS) of EGFR FISH-positive Patients
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Eligible and evaluable participants who were EGFR-FISH positive
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 201 | 199
Months | 9.8 [8.7 to 12.1] | 13.4 [11.5 to 14.8]
Statistical Analysis 1: Comparison: Arm I (Chemo +/- Bevacizumab) vs Arm II (Chemo, Cetuximab, +/- Bevacizumab); Test type: Other; p = 0.054, Log Rank; A stratified log rank test was used; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.66 to 1.00]

4. Secondary Outcome: Progression-Free Survival (PFS) of EGFR FISH-positive Patients by Centralized Review
Description: as for outcome 2
Time Frame: Disease assessment will be repeated every 6 weeks until disease progression while on treatment. After off treatment, the frequency of disease assessment may be reduced to every 3 months until disease progression.
Population: Data are not available for this outcome as central image review was not performed. The study was closed for futility at the interim analysis and therefore there was no need to confirm PFS by central review.
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression-Free Survival (PFS) of the Entire Study Population by Institutional Review
Description: as for outcome 2
Time Frame: as for outcome 4
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 657 | 656
Months | 4.5 [4.2 to 5.1] | 4.6 [4.2 to 5.2]
Statistical Analysis 1: Comparison: Arm I (Chemo +/- Bevacizumab) vs Arm II (Chemo, Cetuximab, +/- Bevacizumab); Test type: Other; p = 0.83, Log Rank; A stratified log rank test was used; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.88 to 1.10]

6. Secondary Outcome: Progression-Free Survival (PFS) of the Entire Study Population by Centralized Review
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 4
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Response Rate (Confirmed Plus Unconfirmed, Complete and Partial Responses) in the Subset of Patients With Measurable Disease in EGFR FISH-positive Patients
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: as for outcome 2
Population: Eligible EGFR FISH positive patients with baseline measurable disease are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 191 | 187
percentage of analyzed participants | 43 [36 to 50] | 47 [39 to 54]
Statistical Analysis 1: Comparison: Arm I (Chemo +/- Bevacizumab) vs Arm II (Chemo, Cetuximab, +/- Bevacizumab); Test type: Other; p = 0.48, Cochran-Mantel-Haenszel; A stratified Cochran-Mantel-Haenszel test was conducted

8. Secondary Outcome: Response Rate (Confirmed Plus Unconfirmed, Complete and Partial Responses) in the Subset of Patients With Measurable Disease in the Entire Study Population
Description: as for outcome 7
Time Frame: as for outcome 2
Population: Eligible patients with baseline measurable disease are included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 623 | 617
percentage of analyzed participants | 36 [33 to 40] | 42 [38 to 46]
Statistical Analysis 1: Comparison: Arm I (Chemo +/- Bevacizumab) vs Arm II (Chemo, Cetuximab, +/- Bevacizumab); Test type: Other; p = 0.060, Cochran-Mantel-Haenszel; A stratified Cochran-Mantel-Haenszel test was conducted

9. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment was evaluated every 3 weeks while one protocol treatment. Chemo and cetuximab is treated for 6 cycles (1 cycle =3 weeks) and Bevacizumab is treated until progression or unacceptable toxicity.
Population: Limited to eligible patients who started treatment, who did not have a major deviation in the treatment protocol, and whose toxicity profile has been completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
Number analyzed (Participants) | 632 | 627
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 5 | 8
  AST, SGOT | 6 | 8
  Acidosis (metabolic or respiratory) | 0 | 1
  Adrenal insufficiency | 0 | 1
  Albumin, serum-low (hypoalbuminemia) | 8 | 7
  Alkaline phosphatase | 2 | 1
  Allergic reaction/hypersensitivity | 9 | 41
  Allergy/Immunology-Other (Specify) | 0 | 2
  Anorexia | 22 | 25
  Apnea | 0 | 1
  Aspiration | 0 | 2
  Ataxia (incoordination) | 1 | 0
  Bilirubin (hyperbilirubinemia) | 2 | 0
  Blood/Bone Marrow-Other (Specify) | 2 | 3
  Bronchospasm, wheezing | 0 | 2
  CNS cerebrovascular ischemia | 2 | 4
  Calcium, serum-high (hypercalcemia) | 2 | 0
  Calcium, serum-low (hypocalcemia) | 1 | 8
  Carbon monoxide diffusion capacity (DL(co)) | 3 | 2
  Cardiac General-Other (Specify) | 2 | 3
  Cardiac troponin I (cTnI) | 0 | 2
  Cardiac-ischemia/infarction | 1 | 1
  Cardiopulmonary arrest, cause unknown (non-fatal) | 1 | 2
  Cognitive disturbance | 1 | 1
  Colitis | 0 | 2
  Colitis, infectious (e.g., Clostridium difficile) | 0 | 1
  Conduction abnormality - Asystole | 1 | 0
  Confusion | 1 | 4
  Constipation | 4 | 4
  Cough | 1 | 2
  Creatinine | 0 | 1
  Cytokine release syndrome/acute infusion reaction | 0 | 10
  Death - Multi-organ failure | 0 | 2
  Death not associated with CTCAE term - Death NOS | 1 | 7
  Dehydration | 27 | 31
  Dermatology/Skin-Other (Specify) | 0 | 3
  Diarrhea | 15 | 19
  Dizziness | 10 | 7
  Dry eye syndrome | 0 | 1
  Dry mouth/salivary gland (xerostomia) | 1 | 0
  Dry skin | 0 | 6
  Dysphagia (difficulty swallowing) | 1 | 2
  Dyspnea (shortness of breath) | 21 | 33
  Edema: limb | 1 | 3
  Encephalopathy | 1 | 0
  Esophagitis | 0 | 2
  Extrapyramidal/involuntary movement/restlessness | 0 | 1
  Eyelid dysfunction | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 74 | 81
  Febrile neutropenia | 27 | 29
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 2 | 0
  GGT (gamma-glutamyl transpeptidase) | 0 | 1
  Gastritis (including bile reflux gastritis) | 0 | 3
  Gastrointestinal-Other (Specify) | 1 | 3
  Glucose, serum-high (hyperglycemia) | 20 | 13
  Glucose, serum-low (hypoglycemia) | 2 | 2
  Heartburn/dyspepsia | 0 | 1
  Hemoglobin | 60 | 48
  Hemolysis | 0 | 3
  Hemorrhage, GI - Abdomen NOS | 0 | 1
  Hemorrhage, GI - Duodenum | 1 | 1
  Hemorrhage, GI - Esophagus | 1 | 0
  Hemorrhage, GI - Jejunum | 0 | 1
  Hemorrhage, GI - Lower GI NOS | 1 | 0
  Hemorrhage, GI - Upper GI NOS | 1 | 2
  Hemorrhage, GI - Varices (esophageal) | 1 | 0
  Hemorrhage, GI - Varices (rectal) | 1 | 0
  Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS | 1 | 1
  Hemorrhage, pulmonary/upper respiratory - Lung | 1 | 3
  Hemorrhage, pulmonary/upper respiratory - Nose | 2 | 1
  Hemorrhage, pulmonary/upper respiratory - Pleura | 1 | 0
  Hemorrhage/Bleeding-Other (Specify) | 1 | 0
  Hiccoughs (hiccups, singultus) | 1 | 1
  Hot flashes/flushes | 1 | 1
  Hypertension | 28 | 17
  Hypotension | 5 | 11
  Hypoxia | 2 | 6
  INR (of prothrombin time) | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 8 | 10
  Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Duodenum | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Esophagus | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 9 | 7
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Pleura | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 1 | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Bladder | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2 | 4
  Inf w/normal ANC or Gr 1-2 neutrophils - Catheter | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Dental | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Joint | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 11 | 8
  Inf w/normal ANC or Gr 1-2 neutrophils - Mucosa | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Pelvis | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Perit cav | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Pleura | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 0 | 5
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 1 | 0
  Infection with unknown ANC - Blood | 1 | 1
  Infection with unknown ANC - Eye NOS | 0 | 1
  Infection with unknown ANC - Lung (pneumonia) | 5 | 3
  Infection with unknown ANC - Sinus | 2 | 0
  Infection with unknown ANC - Skin (cellulitis) | 0 | 1
  Infection with unknown ANC - Upper airway NOS | 0 | 1
  Infection with unknown ANC - Urinary tract NOS | 2 | 1
  Infection with unknown ANC - Wound | 0 | 1
  Infection-Other (Specify) | 4 | 2
  Insomnia | 1 | 5
  Irregular menses (change from baseline) | 0 | 1
  Leukocytes (total WBC) | 74 | 103
  Leukoencephalopathy (radiolographic findings) | 1 | 0
  Local complication - device/prosthesis-related | 0 | 1
  Lymphopenia | 39 | 60
  Magnesium, serum-high (hypermagnesemia) | 0 | 1
  Magnesium, serum-low (hypomagnesemia) | 6 | 28
  Memory impairment | 0 | 1
  Mental status | 0 | 1
  Metabolic/Laboratory-Other (Specify) | 1 | 0
  Mood alteration - anxiety | 0 | 1
  Mood alteration - depression | 3 | 2
  Mucositis/stomatitis (clinical exam) - Esophagus | 1 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2 | 6
  Mucositis/stomatitis (functional/symp) - Oral cav | 0 | 4
  Muscle weakness, not d/t neuropathy - Extrem-lower | 6 | 9
  Muscle weakness, not d/t neuropathy - Extrem-upper | 0 | 1
  Muscle weakness, not d/t neuropathy - Pelvic | 0 | 1
  Muscle weakness, not d/t neuropathy - body/general | 21 | 33
  Nail changes | 0 | 4
  Nasal cavity/paranasal sinus reactions | 0 | 1
  Nausea | 26 | 30
  Neuroendocrine: ADH secretion abnormality | 0 | 2
  Neuropathy: motor | 18 | 10
  Neuropathy: sensory | 57 | 36
  Neutrophils/granulocytes (ANC/AGC) | 158 | 210
  Obstruction, GI - Small bowel NOS | 0 | 1
  Obstruction/stenosis of airway - Bronchus | 1 | 0
  Ocular/Visual-Other (Specify) | 1 | 1
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 1 | 0
  Pain - Abdomen NOS | 5 | 9
  Pain - Back | 1 | 2
  Pain - Bone | 2 | 1
  Pain - Chest wall | 1 | 2
  Pain - Chest/thorax NOS | 1 | 2
  Pain - Extremity-limb | 10 | 12
  Pain - Head/headache | 2 | 1
  Pain - Joint | 19 | 19
  Pain - Muscle | 24 | 14
  Pain - Neck | 1 | 0
  Pain - Neuralgia/peripheral nerve | 1 | 1
  Pain - Oral cavity | 0 | 1
  Pain - Peritoneum | 1 | 0
  Pain - Scrotum | 1 | 0
  Pain - Skin | 0 | 1
  Pain - Stomach | 0 | 1
  Pain-Other (Specify) | 2 | 3
  Pancreatitis | 0 | 1
  Perforation, GI - Colon | 1 | 6
  Perforation, GI - Duodenum | 1 | 0
  Perforation, GI - Small bowel NOS | 0 | 1
  Pericardial effusion (non-malignant) | 0 | 1
  Phosphate, serum-low (hypophosphatemia) | 2 | 8
  Platelets | 51 | 43
  Pleural effusion (non-malignant) | 1 | 0
  Pneumonitis/pulmonary infiltrates | 2 | 8
  Potassium, serum-high (hyperkalemia) | 1 | 4
  Potassium, serum-low (hypokalemia) | 22 | 35
  Proteinuria | 4 | 7
  Pruritus/itching | 0 | 7
  Pulmonary/Upper Respiratory-Other (Specify) | 2 | 2
  Rash/desquamation | 1 | 6
  Rash: acne/acneiform | 0 | 50
  Rash: hand-foot skin reaction | 0 | 4
  Renal failure | 0 | 2
  Renal/Genitourinary-Other (Specify) | 3 | 0
  SVT and nodal arrhythmia - Atrial fibrillation | 2 | 0
  SVT and nodal arrhythmia - Atrial flutter | 1 | 1
  SVT and nodal arrhythmia - SVT tachycardia | 1 | 1
  SVT and nodal arrhythmia - Sinus tachycardia | 1 | 0
  Seizure | 0 | 2
  Sodium, serum-low (hyponatremia) | 29 | 27
  Somnolence/depressed level of consciousness | 1 | 2
  Sudden death | 0 | 1
  Syncope (fainting) | 8 | 7
  Syndromes-Other (Specify) | 0 | 2
  Thrombosis/embolism (vascular access-related) | 0 | 4
  Thrombosis/thrombus/embolism | 26 | 37
  Tinnitus | 0 | 1
  Tremor | 0 | 1
  Tumor lysis syndrome | 0 | 1
  Typhlitis (cecal inflammation) | 1 | 0
  Ulcer, GI - Duodenum | 1 | 1
  Ulcer, GI - Stomach | 0 | 1
  Ulceration | 0 | 1
  Uric acid, serum-high (hyperuricemia) | 1 | 0
  Urticaria (hives, welts, wheals) | 0 | 4
  Ventricular arrhythmia - Ventricular tachycardia | 1 | 0
  Ventricular arrhythmia NOS | 0 | 1
  Visceral arterial ischemia (non-myocardial) | 0 | 1
  Vomiting | 19 | 18
  Weight gain | 0 | 1
  Weight loss | 8 | 4
  Wound complication, non-infectious | 0 | 1

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated every 3 weeks while on protocol treatment. Chemo and cetuximab is treated for 6 cycles (1 cycle =3 weeks) and Bevacizumab is treated until progression, an average of 6 months.
Description: Limited to eligible patients who started treatment, who did not have a major deviation in the treatment protocol, and whose toxicity profile has been completed.
Arm/Group | Arm I (Chemo +/- Bevacizumab) | Arm II (Chemo, Cetuximab, +/- Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 593/657 | 570/656
Serious Adverse Events (participants affected / at risk) | 66/632 | 97/627
Other Adverse Events (participants affected / at risk) | 619/632 | 611/627
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemo +/- Bevacizumab) (N=632) | Arm II (Chemo, Cetuximab, +/- Bevacizumab) (N=627)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 3
Hemoglobin (Blood and lymphatic system disorders) | 2 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Cardiac General-Other (Cardiac disorders) | 3 | 3
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 1
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 | 2
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2 | 0
Ventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 1 | 2
Hemorrhage, GI - Duodenum (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Esophagus (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 | 1
Perforation, GI - Colon (Gastrointestinal disorders) | 0 | 4
Perforation, GI - Duodenum (Gastrointestinal disorders) | 1 | 0
Perforation, GI - Stomach (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 1 | 0
Death - Multi-organ failure (General disorders) | 0 | 2
Death not associated with CTCAE term - Death NOS (General disorders) | 12 | 12
Sudden death (General disorders) | 0 | 1
Syndromes-Other (General disorders) | 1 | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 | 1
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 8
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 0 | 3
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 0 | 5
Inf (clin/microbio) w/Gr 3-4 neuts - Esophagus (Infections and infestations) | 0 | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 2
Infection with unknown ANC - Blood (Infections and infestations) | 2 | 1
Intra-operative Injury-Other (Injury, poisoning and procedural complications) | 1 | 0
Vessel injury-artery - Aorta (Injury, poisoning and procedural complications) | 1 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 1
AST, SGOT (Investigations) | 0 | 1
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 8 | 8
Creatinine (Investigations) | 1 | 0
Leukocytes (total WBC) (Investigations) | 0 | 1
Lymphopenia (Investigations) | 0 | 1
Neuroendocrine: ADH secretion abnormality (Investigations) | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 1
Platelets (Investigations) | 0 | 3
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 | 3
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 17
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 3
Neurology-Other (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage, pulmonary/upper respiratory - Pleura (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Obstruction/stenosis of airway - Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 4 | 4
Visceral arterial ischemia (non-myocardial) (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemo +/- Bevacizumab) (N=632) | Arm II (Chemo, Cetuximab, +/- Bevacizumab) (N=627)
Hemoglobin (Blood and lymphatic system disorders) | 434 | 384
Vision-blurred vision (Eye disorders) | 38 | 33
Constipation (Gastrointestinal disorders) | 261 | 302
Diarrhea (Gastrointestinal disorders) | 195 | 243
Heartburn/dyspepsia (Gastrointestinal disorders) | 70 | 109
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 74 | 162
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 36 | 74
Nausea (Gastrointestinal disorders) | 304 | 318
Pain - Abdomen NOS (Gastrointestinal disorders) | 60 | 86
Vomiting (Gastrointestinal disorders) | 150 | 168
Edema: limb (General disorders) | 80 | 84
Fatigue (asthenia, lethargy, malaise) (General disorders) | 494 | 474
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 56 | 47
Pain - Chest/thorax NOS (General disorders) | 72 | 72
Pain-Other (General disorders) | 63 | 80
Rigors/chills (General disorders) | 49 | 56
Allergic reaction/hypersensitivity (Immune system disorders) | 37 | 90
Infection-Other (Infections and infestations) | 35 | 53
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 82 | 148
AST, SGOT (Investigations) | 81 | 141
Alkaline phosphatase (Investigations) | 138 | 169
Bilirubin (hyperbilirubinemia) (Investigations) | 30 | 32
Creatinine (Investigations) | 52 | 45
Leukocytes (total WBC) (Investigations) | 258 | 289
Lymphopenia (Investigations) | 139 | 166
Metabolic/Laboratory-Other (Investigations) | 39 | 49
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 252 | 305
Platelets (Investigations) | 270 | 233
Weight loss (Investigations) | 163 | 181
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 211 | 244
Anorexia (Metabolism and nutrition disorders) | 245 | 241
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 117 | 179
Dehydration (Metabolism and nutrition disorders) | 104 | 118
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 290 | 266
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 201 | 349
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 34 | 34
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 135 | 200
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 194 | 205
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 56 | 59
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 110 | 122
Pain - Back (Musculoskeletal and connective tissue disorders) | 109 | 126
Pain - Bone (Musculoskeletal and connective tissue disorders) | 50 | 60
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 43 | 38
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 131 | 150
Pain - Joint (Musculoskeletal and connective tissue disorders) | 192 | 194
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 160 | 149
Dizziness (Nervous system disorders) | 129 | 167
Neuropathy: motor (Nervous system disorders) | 62 | 67
Neuropathy: sensory (Nervous system disorders) | 386 | 368
Pain - Head/headache (Nervous system disorders) | 80 | 84
Taste alteration (dysgeusia) (Nervous system disorders) | 131 | 147
Confusion (Psychiatric disorders) | 31 | 40
Insomnia (Psychiatric disorders) | 95 | 131
Mood alteration - anxiety (Psychiatric disorders) | 61 | 70
Mood alteration - depression (Psychiatric disorders) | 58 | 60
Proteinuria (Renal and urinary disorders) | 36 | 50
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 48 | 66
Cough (Respiratory, thoracic and mediastinal disorders) | 239 | 248
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 285 | 290
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 86 | 115
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 23 | 38
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 40 | 37
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 17 | 82
Dry skin (Skin and subcutaneous tissue disorders) | 64 | 220
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 315 | 293
Nail changes (Skin and subcutaneous tissue disorders) | 37 | 67
Pruritus/itching (Skin and subcutaneous tissue disorders) | 49 | 122
Rash/desquamation (Skin and subcutaneous tissue disorders) | 42 | 155
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 40 | 425
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 | 54
Hypertension (Vascular disorders) | 124 | 96
Hypotension (Vascular disorders) | 55 | 79
Thrombosis/thrombus/embolism (Vascular disorders) | 54 | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT00946712/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT00946712/ICF_001.pdf